CLINICAL TRIAL: NCT02017990
Title: The Levels of Marine n-3 Polyunsaturated Fatty Acids in Plasma Phospholipids as a Prognostic Marker of Mortality and Graft Loss Endpoints in Renal Transplant Recipients.
Brief Title: Plasma Marine n-3 Polyunsaturated Fatty Acids and Patient and Graft Survival
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: REK 2012/1419
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Disorder of Transplanted Kidney
Keywords: Renal transplantation; n-3 polyunsaturated fatty acids; Mortality; Graft loss; Rejection
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma phospholipids.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Renal transplant recipients: No intervention. Measurements of plasma marine n-3 polyunsaturated fatty acids levels, indicating intake of fish and seafood.

SUMMARY:
This study will evaluate the association between n-3 polyunsaturated fatty acids and patient and graft survival. The association between other fatty acids and mortality and graft loss endpoints will also be evaluated.

DETAILED DESCRIPTION:
This observational study focuses on the effects of marine n-3 polyunsaturated fatty acids (PUFAs) intake, measured as fatty acid levels in plasma phospholipids, and mortality and graft loss endpoints in renal transplant recipients. Data on morbidity, mortality and graft loss in The Norwegian Renal Registry is matched against data on fatty acid composition in a large renal transplantation cohort of approximately 2000 patients with a median follow up time of about 5 years. It is a follow up study, although retrospectively evaluated. It will evaluate the role of marine n-3 PUFAs as a prognostic marker in renal transplantation by investigating the association between the levels (weight percentage of total fatty acids) of marine n-3 PUFAs in plasma phospholipids and events, including mortality and graft loss.

ELIGIBILITY:
Inclusion Criteria:

* Received a renal transplant. Signed informed consent.

Exclusion Criteria:

* Under the age of 16 years.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Renal transplant recipients
Sampling Method: Probability Sample
Enrollment: 2002 (Actual)
Dates: Start 1999-10; Primary Completion 2012-08 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | Up to 12 years.
  First patient recruited October 1999 and all remaining patients were censored at August 2012.

SECONDARY OUTCOMES:
Loss of function in the renal transplant. | Up to 12 years.
  As for primary endpoint.

OTHER OUTCOMES:
Cause specific mortality rates. | Up to 12 years.
  As for the primary endpoint. Mortality rates for cardiac, cerebrovascular, infectious disease and malignancies.
Cause specific graft loss. | Up to 12 years.
  As for the primary endpoints. Graft loss rates for rejection and recurrence as well as total and death censored graft loss will be registered.
Rejection rate. | Up to 12 years.
  As for the primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Ivar Eide, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Rikshospitalet, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Eide IA, Jenssen T, Hartmann A, Diep LM, Dahle DO, Reisaeter AV, Bjerve KS, Christensen JH, Schmidt EB, Svensson M. The association between marine n-3 polyunsaturated fatty acid levels and survival after renal transplantation. Clin J Am Soc Nephrol. 2015 Jul 7;10(7):1246-56. doi: 10.2215/CJN.11931214. Epub 2015 Jun 10. PMID 26063768